CLINICAL TRIAL: NCT01128400
Title: Inhibition of Lipolysis in Oral Cavity and Fat Perception in Humans
Brief Title: Fat Perception in Humans (09-0873)
Acronym: OT
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 09-0873
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Obesity
Keywords: obesity; orlistat; taste perception
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood will be collected and frozen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- rs1761667- AA genotype: subjects carrying the CD36 genotype rs1761667, i.e. a Single Nucleotide Polymorphism that significantly reduces CD36 level and has a minor allele frequency of 38-48%.
- rs1761667-GG genotype: subjects who are homozygous of CD36 genotype rs1761667-G allele.
- rs1761667-AG genotype: Heterozygous of CD36 gene rs1761667-A genotype.

SUMMARY:
There are many substances naturally present in the mouth that may help us taste fat in food. Two of these substances (lipases and CD36) will be examined in this study.

The presence of fat in food increases food tastiness, therefore people often over-eat high-fat foods and gain weight. The purpose of this study is to determine if blocking lipases and some genetic variations in the CD36 gene will make fatty food less tasty so that people eat less. Our hypothesis is that Orlistat and a particular gene will increase one's ability to detect fat.

DETAILED DESCRIPTION:
1. Determine the effect of lipolysis inhibition in oral cavity on orosensory detection of fat in humans.

   Hypothesis: Orally applied Orlistat will increase detection thresholds of TAGs but not FFA in humans.

   To test this hypothesis we will measure triolein (a TAG) and oleic acid (a FFA) taste detection thresholds with a three-alternative forced-choice (3-AFC) ascending concentration method under two conditions (Orlistat day vs. Control day). To control for olfactory input, subjects will be assessed wearing noseclips.
2. Determine the effect of CD36 variants on fat taste perception in humans. Hypothesis: SNPs that associate with reduced CD36 expression will be associated with higher FFA and TAG detection thresholds

To test this hypothesis we will measure triolein and oleic acid taste detection thresholds in subjects who carry of the common CD36 e-SNP rs1761667 (i.e. a SNP that significantly reduces CD36 level and has a minor allele frequency of 38-48%). We expect subjects who are at least heterozygous for the expression reducing allele to have higher triolein and oleic acid taste detection thresholds compared to non-carrier subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index greater than 30 kg/m²

Exclusion Criteria:

* smokers or who quit smoking less than six months ago
* pregnancy
* breastfeeding
* diabetes
* taking medications that might affect taste perception
* previous malabsorptive or restrictive intestinal surgery

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 40 obese subjects will participate in this study. Subjects will be men and women and will include all races and ethnic groups. The two groups (carriers and non-will be matched as closely as possible in age, sex, body mass index (kg/m²) and race distributions.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Y Pepino de Gruev, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: May 2010- August 2011 recruited by local posters and media advertising via the Washington University Research Participant Registry.
Pre-assignment Details: 40 subjects signed consent form and were screened for rs1761667 genotype and three groups (i.e., AA, AG and GG) matched in age and BMI were invited to participate on the taste test.
Period: Overall Study
Arm/Group | rs1761667- AA Genotype | rs1761667-GG Genotype | rs1761667-AG Genotype
Started | 8 | 9 | 23
Completed | 6 | 8 | 7
Not Completed | 2 | 1 | 16
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Screening failure | 1 | 0 | 0
Not completed — were not invited to participate on taste | 0 | 0 | 15
Not completed — Excluded due to sinus problems | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Three groups of obese subjects (body mass index [BMI] >30 kg/m2) participated in this study. The three groups were matched on age, because there is a generic decline in taste perception with age.
Groups:
- rs1761667- AA Genotype: Obese subjects carrying the CD36 genotype rs1761667, i.e. a Single Nucleotide Polymorphism that significantly reduces CD36 level
- rs1761667-GG Genotype: Obese subjects who are homozygous of CD36 genotype rs1761667-G allele.
- rs1761667-AG Genotype: Obese subjects who are heterozygous of CD36 gene rs1761667-A genotype.
- Total: Total of all reporting groups
Arm/Group | rs1761667- AA Genotype | rs1761667-GG Genotype | rs1761667-AG Genotype | Total
Number analyzed (Participants) | 6 | 8 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (14.0) | 39.1 (7.0) | 39.6 (6.4) | 39.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 18
  Male | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Oleic Acid Detection Level
Description: We will measure oleic acid detection levels as a marker of subjects' ability to detect free fatty acids. Oleic acid taste detection thresholds were separately assessed using a three-alternative forced-choice (i.e. 3-AFC) ascending concentration.
Time Frame: Ranges from 5 days after screening to several weeks, pending availablity of participant.
Measure: Mean (Standard Error); unit: log10 (%W/V OLEIC ACID)
Arm/Group | rs1761667- AA Genotype | rs1761667-GG Genotype | rs1761667-AG Genotype
Number analyzed (Participants) | 6 | 8 | 7
log10 (%W/V OLEIC ACID) | -0.3 (0.3) | -1.2 (0.2) | -1.0 (0.3)
Statistical Analysis 1: Comparison: rs1761667- AA Genotype vs rs1761667-GG Genotype vs rs1761667-AG Genotype; Test type: Superiority or Other; p = 0.05, ANOVA

2. Primary Outcome: Triolein Detection
Description: We will measure triolein detection levels as a marker of subjects' ability to detect triglyceride. Triolein taste detection thresholds were separately assessed using a three-alternative forced-choice (i.e. 3-AFC) ascending concentration.
Time Frame: Ranges from 5 days after screening to several weeks, pending availablity of participant.
Measure: Mean (Standard Error); unit: log10 (%W/V TRIOLEIN)
Arm/Group | rs1761667- AA Genotype | rs1761667-GG Genotype | rs1761667-AG Genotype
Number analyzed (Participants) | 6 | 8 | 7
log10 (%W/V TRIOLEIN) | 0.55 (0.25) | -0.33 (0.22) | -0.04 (0.23)
Statistical Analysis 1: Comparison: rs1761667- AA Genotype vs rs1761667-GG Genotype vs rs1761667-AG Genotype; Test type: Superiority or Other; p = 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 2 year
Description: For the taste testing study, all taste testing stimuli were prepared in a metabolic kitchen using proper food safety guidelinse and none of the stimuli that were tasted were swallowed (i.e. we used a sip and spit technique). Therefore, we did not anticipate and did not planned on collecting/assessing adverse events.
Arm/Group | rs1761667- AA Genotype | rs1761667-GG Genotype | rs1761667-AG Genotype
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No